CLINICAL TRIAL: NCT05596409
Title: ELACESTRANT in Women and Men With CDK4/6 Inhibitor-Naive Estrogen Receptor Positive, HER-2 Negative Metastatic Breast Cancer: An Open-Label Multicenter Phase 2 Study (ELCIN)
Brief Title: ELACESTRANT in Women and Men With CDK4/6 Inhibitor-Naive Estrogen Receptor Positive, HER-2 Negative Metastatic Breast Cancer Study
Acronym: ELCIN
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Stemline Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STML-ELA-0322
Record Dates: First submitted 2022-10-24; First posted 2022-10-27 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Metastatic Breast Cancer
Keywords: metastatic breast cancer; breast cancer; elacestrant
MeSH Terms: conditions — Breast Neoplasms | interventions — elacestrant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Elacestrant (Experimental): Subjects will take a starting dose of 400 mg of elacestrant dihydrochloride in tablet form once daily for up to 6 months.
  Interventions: Drug: Elacestrant

INTERVENTIONS:
Drug: Elacestrant — Starting dose 400 mg elacestrant dihydrochloride administered orally once daily for an estimated 6 months of treatment.

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of elacestrant over the course of 6 months in patients with estrogen receptor positive (ER+)/human epidermal growth factor receptor-2 negative (HER2-) advanced/metastatic breast cancer who received no prior cyclin-dependent kinase targeting enzymes CDK4 and CDK6 inhibitor (CDK4/6i) in the metastatic setting.

DETAILED DESCRIPTION:
This is a Phase 2 trial evaluating the efficacy of elacestrant in patients with ER+/HER2- advanced/metastatic breast cancer who received one or two prior hormonal therapies and no prior CDK4/6i in the metastatic setting.

The study duration for each patient is estimated to be:

* Screening Phase: Up to 28 days prior to Cycle 1, Day 1 (C1D1);
* Treatment Phase: From C1D1 until the date of radiologically documented progression, or treatment discontinuation due to other reasons.
* Survival Follow-Up Phase: All patients will be followed for survival approximately every 3 months up to 24 months after enrollment of the last patient.

Patients will be followed for adverse events (AEs) for 28 days after the last treatment administration.

ELIGIBILITY:
Inclusion Criteria:

1. Patient has signed the informed consent before all study specific activities are conducted.
2. Women or men aged ≥18 years (or the minimum age of consent as per local law), at the time of informed consent signature. Female patients may be either postmenopausal or premenopausal/perimenopausal.

   1. Premenopausal or perimenopausal women and men must be concurrently given a luteinizing hormone-releasing hormone (LHRH) agonist starting at least 4 weeks before the start of trial therapy and is planning to continue LHRH during the study.
   2. For perimenopausal women to be considered of non-childbearing potential, follicle-stimulating hormone (FSH) levels must be >40 milli-international units per milliliter (mIU/mL).
3. Documentation of histopathologically or cytologically confirmed ER+, HER2-breast cancer, per local laboratory, as per the American Society of Clinical Oncology (ASCO)/College of American Pathologists (CAP) guidelines. Note: In the context of this trial, ER status will be considered positive if ≥10% of tumor cells demonstrate positive nuclear staining by immunohistochemistry.
4. Radiological disease progression during or after the most recent therapy in the advanced/metastatic setting
5. Patient has received at least one (and up to two) prior hormonal therapy in the advanced/metastatic setting.
6. Patients with disease relapse while on adjuvant endocrine therapy after the 2 first years, or with disease relapse within 12 months of completing adjuvant endocrine therapy are allowed (i.e., patients with secondary-resistant breast cancer according to the 5th European School of Oncology (ESO)-European Society for Medical Oncology (ESMO) international consensus guidelines for advanced breast cancer, Cardoso et al 2020). This therapy will be considered as first line treatment for eligibility purposes.
7. At least one measurable lesion as per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 or a mainly lytic bone lesion for bone only disease.
8. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
9. Patient has adequate bone marrow and organ function, as defined by the following laboratory values:

   1. Absolute neutrophil count (ANC) ≥1.5 × 10^9/liter(L)
   2. Platelets ≥100 × 10^9/L
   3. Hemoglobin ≥9.0 grams(g)/deciliter(dL)
   4. Potassium, sodium, calcium (corrected for serum albumin) and magnesium, Common Terminology Criteria for Adverse Events (CTCAE) v5.0 grade ≤1. Note: Corrected calcium for serum albumin must be calculated manually by the site using the Payne formula: Corrected calcium (milligrams [mg]/dL) = measured total calcium (mg/dL) + 0.8 (Normal albumin [g/dL] - serum albumin [g/dL]), where normal albumin is usually defaulted to 4.0 g/dL.
   5. Cockcroft-Gault based creatinine clearance ≥50 milliliters per minute (mL/min). Note: Creatinine clearance (male) = ([140-age in years] × weight in kilograms [kg])/ ([serum creatinine in mg/dL] × 72) Creatinine clearance (female) = (0.85 × [140-age in years] × weight in kg)/ ([serum creatinine in mg/dL] × 72)
   6. Serum albumin ≥3.0 g/dL (≥30 g/L)
   7. In absence of liver metastases, alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤3.0 × upper limit of normal (ULN). If the patient has liver metastases, ALT and AST ≤5 × ULN
   8. If the patient has liver metastases, ALT, and AST ≤5.0 × ULN
   9. Total serum bilirubin <1.5 × ULN except for patients with Gilbert's syndrome who may be included if the total serum bilirubin is ≤3.0 × ULN or direct bilirubin ≤ 1.5 × ULN. Note: Laboratory assessments may be repeated during the Screening Phase after supplementation or transfusions (a single red blood cells transfusion is allowed once during the screening period).

Exclusion Criteria:

1. Active or newly diagnosed central nervous system (CNS) metastases, including meningeal carcinomatosis.
2. Patients with advanced, symptomatic visceral crisis who are at risk of life-threatening complications in the short term, including massive uncontrolled effusions (peritoneal, pleural, pericardial) and liver involvement of >50%.
3. Prior chemotherapy, elacestrant, or CDK4/6i in the advanced/metastatic setting.
4. Patients with only disease relapse while on the first 2 years of adjuvant endocrine therapy i.e., patients with primary endocrine resistance, are not eligible.
5. Patient has a concurrent malignancy or history of invasive malignancy within 3 years of enrollment, with the exception of basal or squamous cell skin cancer, superficial bladder cancer, or carcinoma in situ of the cervix that has completed curative treatment.
6. Uncontrolled significant active infections.

   1. Patients with hepatitis B virus (HBV) and/or hepatitis C virus (HCV) infection must have undetectable viral load during screening.
   2. Patients known to be human immunodeficiency virus (HIV)+ are allowed as long as they have undetectable viral load at baseline.
7. Major surgery within 28 days before starting trial therapy.
8. Systemic radiotherapy within 14 days before starting trial therapy, or central nervous system (CNS) radiotherapy within 28 days before starting trial therapy. Inability to take oral medication, refractory or chronic nausea, gastrointestinal condition (including significant gastric or bowel resection), history of malabsorption syndrome, or any other uncontrolled gastrointestinal condition that may impact the absorption of study drug.
9. Known intolerance to elacestrant or any of its excipients.
10. Females of childbearing potential who do not agree to use a highly effective method of contraception and to abstain from donating/freezing ova within 28 days of the first dose of study treatment through 120 days after the last dose of study treatment. Highly effective non-hormonal methods of contraception should be used.
11. Men who do not agree to abstain from donating/freezing sperm, or to use a highly effective method of contraception within 28 days of the first dose of study treatment through 120 days after the last dose of study treatment. For subjects (who have not undergone vasectomy) with female partners of childbearing potential, the subject and his partner must use highly effective methods of contraception.
12. Females who are pregnant or breastfeeding. Females should not get pregnant during study treatment and for 120 days after last dose of study treatment. Females should not breastfeed during administration of elacestrant and for 1 week after receiving the last dose.
13. Patient is currently receiving or received any of the following medications prior to first dose of trial therapy:

    1. Investigational anti-cancer therapy within 14 days (28 days in case of anticancer antibody-based treatments) or 5 half-lives, whichever is shorter.
    2. Fulvestrant treatment (last injection) <42 days before first dose of study drug.
    3. Any other endocrine therapy <14 days before first dose of study drug.
    4. Known strong or moderate inducers or inhibitors of cytochrome P450 (CYP) 3A4 within 14 days or 5 half-lives, whichever is shorter.
    5. Herbal preparations/medications within 7 days. These include, but are not limited to, St. John's wort, kava, ephedra (ma huang), gingko biloba, dehydroepiandrosterone (DHEA), yohimbe, saw palmetto, and ginseng.
14. Any severe medical or psychiatric condition that in the opinion of the investigator(s) would preclude the patient's participation in a clinical study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2023-05-19 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | 36 months
  PFS is defined as time from the date of the first dose to the date of the first radiological documentation of disease progression or death, whichever comes first.

SECONDARY OUTCOMES:
Overall response rate | 24 months
  Proportion of patients who achieve a best overall response of partial response or complete response
Duration of response | 36 months
  Time from the date of first documented complete response or partial response until the first radiological documentation of disease progression or death, whichever comes first
Clinical benefit rate | 36 months
  Proportion of patients who achieve a best overall response of confirmed complete response or partial response or durable stable disease (duration at least 24 weeks from date of first dose)
Overall survival | 36 months
  Time from the date of the first dose to the date of the first radiological documentation of disease progression or death, whichever comes first

CONTACTS AND LOCATIONS:
Locations (34):
- United States (11):
  - Highlands Oncology Group, PA, Springdale, Arkansas
  - OPN Healthcare, Arcadia, California
  - University of Colorado Cancer Center, Aurora, Colorado
  - Morton Plant Hospital - Baycare Health System, Clearwater, Florida
  - Northwestern University, Northwestern Feinberg School of Medicine Prentice Women's Hospital, Chicago, Illinois
  - Inventa Center for Cancer Research at Fort Wayne Medical Oncology and Hematology, Fort Wayne, Indiana
  - Alliance for Multispecialty Research, Merriam, Kansas
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - The Toledo Clinic, Toledo, Ohio
  - UT Health San Antonio Mays Cancer Center, San Antonio, Texas
  - Quality Cancer Care Alliance (QCCA) Northwest Medical Specialties, Tacoma, Washington
- Brazil (8):
  - Centro de Pesquisas Clinicas em Oncologia (Center for Clinical Research in Oncology (CPCO)) - Hospital Evangélico de Cachoeiro de Itapemirim, Cachoeiro de Itapemirim, Espírito Santo
  - Hospital São Lucas PUCRS - Centro de Pesquisa em Oncologia (CPO), Porto Alegre, Rio Granda Do Sul
  - Hospital de Clinicas de Porto Alegre, Porto Alegre, Rio Granda Do Sul
  - Centro de Pesquisas Oncologicas, Florianópolis, Santa Catarina
  - Hospital de Amor de Barretos, Barretos, São Paulo
  - Centro de Estudos e Pesquisas de Hematologia e Oncologia- CEPHO, Santo André, São Paulo
  - Centro De Pesquisa Clinica DO Hospital Sirio-Libanes - UNIDADE Brasilia, Brasília
  - Clinica de Pesquisas e Centro de Estudos Em Oncologia Ginecologica e Mamaria Ltda, São Paulo
- Bulgaria (3):
  - Complex Oncology Center, Plovdiv
  - COMPLEX ONCOLOGICAL CENTER - Shumen, Shumen
  - COC Veliko Tarnovo, Veliko Tarnovo
- Georgia (6):
  - Cancer Research Centre, Tbilisi
  - Innova Medical Center, Tbilisi
  - LTD Simon Khechinashvili University Clinic, Tbilisi
  - Multiprofile Clinic Consilium Medulla, Tbilisi
  - Institute of Clinical Oncology, Tbilisi
  - Todua Clinic, Tbilisi
- Mexico (4):
  - I CAN Oncology Center, Centro Medico AVE, Monterrey, Nuevo León
  - Torre Medica Hospital Dalinde, Mexico City
  - Fucam, Ac., Mexico City
  - Unidad Médica Onco-Hematológica, Puebla City
- Romania (2):
  - Institutul Oncologic "Prof. Dr. Ion Chiricuta" Cluj Napoca, Cluj-Napoca, Cluj
  - Centrul de Oncologie "Sf. Nectarie", Craiova, Dolj